CLINICAL TRIAL: NCT04704024
Title: A Phase III, Randomized, 2x2 Factorial Trial to Assess the Efficacy of Antiviral Therapy in Women and Infants in Reducing Vertical Transmission of Hepatitis B in Africa
Brief Title: Reducing Vertical Transmission of Hepatitis B in Africa
Acronym: REVERT-B
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jodie A. Dionne, MD, Associate Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-300006586; 5R01HD101545 (NIH)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Hepatitis B Infection
Keywords: perinatal infection, hepatitis B in pregnancy
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; Lamivudine

STUDY DESIGN:
Intervention Model Description: 2x2 factorial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pregnant women will be randomized in open label fashion to early or late initiation of TDF.
  Infants will be randomized to receive lamivudine or matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregnant Women - Tenofovir (Experimental): Women will be randomized to early initiation (enrollment at 14-28 weeks pregnant) vs standard initiation (at 28 weeks pregnant) of tenofovir disoproxil fumarate (TDF) 300 mg daily oral medication until delivery.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- Newborn Infants - Lamivudine (Placebo Comparator): Infants exposed to HBV at birth will be randomized to receive oral lamivudine post-exposure prophylaxis or matching placebo. Medication will be administered twice daily for 6 months.
  Interventions: Drug: Lamivudine Oral Solution

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — oral TDF medication 300 mg daily
  Other Names: TDF
  Arms: Pregnant Women - Tenofovir
Drug: Lamivudine Oral Solution — Oral lamivudine with weight-based dosing BID from birth until 6 months of age
  Other Names: 3TC
  Arms: Newborn Infants - Lamivudine

SUMMARY:
Hepatitis B virus is an infection that can be easily transmitted from women to newborns at the time of delivery. Our objective is to identify novel options that are effective and safe in preventing perinatal transmission of hepatitis B in Africa. The REVERT-B study (Reducing Vertical Transmission of Hepatitis B in Africa) is a clinical trial designed to test a new strategy of using antiviral medication in high-risk pregnant women and newborns to reduce the risk of hepatitis B transmission. The study will measure efficacy, safety, tolerability and adherence to medication.

DETAILED DESCRIPTION:
The REVERT-B trial is a multi-center, phase III, randomized 2x2 factorial study designed to test the efficacy of early maternal TDF vs standard duration and neonatal 3TC prophylaxis compared to matching placebo in preventing HBV MTCT. Eligible pregnant women with HBV in prenatal care (n=450) will be randomized 1:1:1:1 to one of four maternal and neonatal prophylaxis combinations (shown as A-D in the figure below). Women will initiate daily oral TDF early (2nd trimester) or at the standard time per WHO guidelines (3rd trimester) and will continue TDF until delivery. The current WHO standard of care in pregnant women with HBV (EAg+) in Cameroon is TDF prophylaxis from 28 weeks until delivery. Newborns will receive liquid 3TC or matching placebo for the first six months of life to provide coverage until the vaccine series is complete. All infants in the study will be offered the 4-dose HBV vaccine series starting at birth.

The 2x2 factorial design allows for two simultaneous studies where we first assess efficacy of early maternal prophylaxis (Aim 1) and secondarily assess efficacy of neonatal prophylaxis (Aim 2). The study endpoint for both aims is the MTCT rate (proportion of infants HBsAg+) at 6-9 months of age. Women and infants will be followed until 6-9 months after delivery and subaims will assess safety and adherence to maternal TDF and neonatal 3TC. Plasma testing will be used to measure medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* prenatal clinic patient,
* age ≥16 years,
* 14-32 weeks gestational age according to clinic dating based on LMP or ultrasound,
* active hepatitis B with risk of vertical transmission (HBsAg+ AND HBeAg+ or HBV DNA >1000 IU/ML),
* plan to receive follow up care and deliver at study facility,
* capable of providing informed consent.

Exclusion Criteria:

* HIV positive (according to HIV antibody testing performed at the initial prenatal visit)
* known liver cirrhosis or end-stage liver disease,
* elevated liver enzymes (ALT >5x upper limit of normal),
* elevated serum creatinine (>1.4 mg/dl)
* currently taking tenofovir medication
* allergy or intolerance to tenofovir study medication,
* known fetal anomaly in the current pregnancy,
* clinical illness requiring hospitalization at the time of enrollment
* evidence of early labor at the time of enrollment.

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — eligible if pregnant
Enrollment: 450 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Vertical Transmission of hepatitis B Infection | 6-9 months of age
  The proportion of infants with Hepatitis B surface antigen positivity (SAg+)
Virologic Suppression | at delivery
  The proportion of women with a suppressed HBV DNA viral load (<10 IU/mL).

SECONDARY OUTCOMES:
In utero HBV infection | at birth
  HBV infection (SAg+, PCR positive)
Maternal Adherence to TDF | 8 weeks after starting medication
  HPLC measurement of serum
Maternal Adherence to TDF | at delivery
  HPLC measurement of serum
Infant Adherence to 3TC | 12 weeks after starting 3TC
  HPLC measurement of serum
Infant Adherence to 3TC | 24 weeks after starting 3TC
  HPLC measurement of serum
Hepatitis B Flare | 12 weeks after delivery
  Increase in ALT (>2x ULN) after stopping TDF at delivery
Hepatitis B Flare | 24 weeks after delivery
  Increase in ALT (>2x ULN) after stopping TDF at delivery
Preterm delivery | assessed at delivery
  Delivery <37 weeks gestational age
Composite Adverse Birth Outcomes | during pregnancy or up to 28 days after delivery
  PTD, SAB, IUFD, neonatal death
Incident HIV infection during pregnancy | at delivery
  Maternal HIV infection with seroconversion to positive test
Retention in Prenatal Care | assessed at time of delivery
  at least 4 ANC visits after 28 weeks GA

CONTACTS AND LOCATIONS:
Overall Officials: Jodie Dionne, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States